CLINICAL TRIAL: NCT04588961
Title: Comparison of Trapeziectomy With Suspensionplasty and Carpometacarpal Joint Replacement in Treatment of Basal Thumb Osteoarthritis: Randomised Clinical Trial
Brief Title: Trapeziectomy Suspensionplasty Versus Carpometacarpal Joint Replacement in Treatment of Basal Thumb Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WarsawMU/thumb
Record Dates: First submitted 2020-09-25; First posted 2020-10-19 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-09

CONDITIONS: Carpometacarpal Osteoarthritis; Rhizarthrosis; Thumb Osteoarthritis
Keywords: Thumb; Osteoarthritis; Trapeziectomy; Alloplasty; Biomechanics
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement

STUDY DESIGN:
Intervention Model Description: Patients would be assigned randomly to 2 different groups
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will not be informed which type of prosthesis was used in particular patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Patients undergoing trapeziectomy with suspensionplasty for primary basal thumb osteoarthritis
  Interventions: Procedure: Trapeziectomy with suspensionplasty
- Study group (Active Comparator): Patients undergoing joint alloplasty using prothesis for primary basal thumb osteoarthritis
  Interventions: Procedure: Joint alloplasty

INTERVENTIONS:
Procedure: Trapeziectomy with suspensionplasty — Surgical removal of trapezium bone and ligamentoplasty of first metacarpal bone using abductor pollicis tendon
  Arms: Control group
Procedure: Joint alloplasty — Surgical removal of degenerated joint surfaces nad replacement using modern designed prothesis
  Other Names: Joint replacement
  Arms: Study group

SUMMARY:
This study compares and evaluates differences in movement analysis, patient-reported outcome, radiological assesment and muscular function between patients undergoing carpometacarpal joint arthroplasty with use of modern implants and trapeziectomy with suspensionplasty

DETAILED DESCRIPTION:
Osteoarthritis of first carpometacarpal joint is the most common degenerative disease of upper limb. According to data available in literature, it affects about 30% of women and 6% of men at the age of 45. Increasing with age, it rises up to 90% in people by the age of 80. Due to more widely spread electronic devices in offices, at work, at home which requires usage of thumb, increase in numbers mentioned above is strongly probable. The main symptoms are: pain, loose of grip strength and loose of function. The latter is most important fact, since about 50% of hand function is possible only with healthy thumb.

In many cases osteoarthritis can be treated by combined NSAIDs and splinting with rehabilitation. Sometimes when symptoms do not respond to non-operative treatment, there is a need for surgery. Trapeziectomy is the most common choice for operative treatment for end-stage basal thumb osteoarthritis. However, many other techniques were developed, there is continuous dispute over selecting the optimal . One of the most promising is arthroplasty using prosthesis. Last years many important advances were made in a design of implant and materials. Moreover the investigators now have many longer outcomes of such operation made in the past. All this data make us think more about using this technique often, since there are papers which show superiority over classical trapeziectomy. Even though there are several studies comparing functional and objective outcome of those techniques, there is a lack of evidence in terms of biomechanical analysis, thenar muscle activity and changes in movement patterns. Moreover there is no study published so far which considers modern implants and trapeziectomy with suspensionplasty. The aim of the study is to examine relationships between movement analysis (kinematic and functional outcomes), patient reported outcome measures (PROMS) and X-ray measurement, electromyography both pre- and post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of carpometacarpal joint III or III/IV in Eaton classification assessed by two different radiologists
* symptoms that do not respond to non-operative treatment for 8 weeks
* no counterindications for anaesthesia
* signed agreement for taking a part into trial

Exclusion Criteria:

* patient do not agree to take a part into study
* problems with communication with patient
* unstable cardiac disease
* reoperations
* previous surgical interventions in hand
* neuro-muscular diseases
* rheumatological background of disease
* diagnosed cervical spine disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in patients reported outcomes - DASH (Disabilities of Arm, Shoulder and Hand) | at baseline, 6 weeks and 6 months postoperatively
  To measure overall disabilities of upper limb. Results range from 0 to 100, with lower scores corresponding to better outcomes.

SECONDARY OUTCOMES:
Changes in patients reported outcomes - PRWE (Patient Related Wrist Evaluation) | at baseline, 6 weeks and 6 months postoperatively
  To measure wrist pain and disability in activities of daily living. Results range from 0 to 50, with lower scores corresponding to better outcomes.
Changes in patients reported outcomes - Michigan Hand Outcomes Questionaire | at baseline, 6 weeks and 6 months postoperatively
  To explore differences in higher levels of activity at work and social participation. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients reported outcomes - SF-36 (Short Form 36) | at baseline, 6 weeks and 6 months postoperatively
  To explore differences in quality of life. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients reported outcome measures - VAS (Visual Analogue Score) | at baseline, 6 weeks and 6 months postoperatively
  To explore differences in pain. Results range from 0 to 100, with lower scores corresponding to better outcomes.
Changes in carpometacarpal, carpophalangeal and wrist range of motion | at baseline, 6 weeks and 6 months postoperatively
  To explore differences in range of motion. This parameter will be measured with goniometer in flexion, extension, adduction and abduction in all thumb joints. Outcomes would be numers of degrees ranging from 0-360, with higher number corresponding with better outcomes
Changes in usage of painkillers | at baseline, 6 weeks and 6 months postoperatively
  To asses evolution of post-operative thumb pain. Dosage, frequency of utilisation and type of medicines will be measured in self-designed questionnaire, with lower dosage, lower frequency and less powerful medicines corresponding with better results
Operation related complications | at baseline, 6 weeks and 6 months postoperatively
  To count and asses all complications that may occur during surgery and in postoperative period
Arthroplasty revision surgeries | at baseline, 6 weeks and 6 months postoperatively
  To count and asses the reason of all revision surgeries that may occur during postoperative period
Biomechanical 3D motion analysis | at baseline, 6 weeks and 6 months postoperatively
  Movements in whole range are measured using 3D motion analysis, using a special software. With more physiological movement patterns corresponding with better results
Radiological outcome on x-rays | at baseline, 6 weeks and 6 months postoperatively
  To asses any changes in alignment of implants with would be measured with degrees (angles) with more degrees of change after operation corresponding with worse outcome
Muscle strength outcomes | at baseline, 6 weeks and 6 months postoperatively
  Muscle strength during grip measured using maximal voluntary isometric contraction (MVIC)
EMG measured bioelectrical potentials | at baseline, 6 weeks and 6 months postoperatively
  Percutaneus electromyography (EMG) will be performed to measure bioelectrical potentials of thumb muscles, to assess ability to contracture

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Stępiński, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
It is still undecided because number of researchers included in the study is unknown

REFERENCES:
- [Background] Sodha S, Ring D, Zurakowski D, Jupiter JB. Prevalence of osteoarthrosis of the trapeziometacarpal joint. J Bone Joint Surg Am. 2005 Dec;87(12):2614-2618. doi: 10.2106/JBJS.E.00104. PMID 16322609
- [Background] Deiler S. [Basal joint osteoarthritis of the thumb]. Orthopade. 2019 Apr;48(4):351-366. doi: 10.1007/s00132-019-03707-8. German. PMID 30843103
- [Background] Weiss AC, Goodman AD. Thumb Basal Joint Arthritis. J Am Acad Orthop Surg. 2018 Aug 15;26(16):562-571. doi: 10.5435/JAAOS-D-17-00374. PMID 29969109
- [Background] Wajon A, Vinycomb T, Carr E, Edmunds I, Ada L. Surgery for thumb (trapeziometacarpal joint) osteoarthritis. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD004631. doi: 10.1002/14651858.CD004631.pub4. PMID 25702783
- [Background] Mahoney JD, Meals RA. Trapeziectomy. Hand Clin. 2006 May;22(2):165-9. doi: 10.1016/j.hcl.2006.02.003. PMID 16701128
- [Background] Naram A, Lyons K, Rothkopf DM, Calkins ER, Breen T, Jones M, Shufflebarger JV. Increased Complications in Trapeziectomy With Ligament Reconstruction and Tendon Interposition Compared With Trapeziectomy Alone. Hand (N Y). 2016 Mar;11(1):78-82. doi: 10.1177/1558944715617215. Epub 2016 Jan 14. PMID 27418894
- [Background] Sivakumar BS, Graham DJ. APL Lasso Suspensionplasty for Trapeziectomy. Tech Hand Up Extrem Surg. 2020 Sep;24(3):108-113. doi: 10.1097/BTH.0000000000000276. PMID 31876776
- [Background] Wang T, Zhao G, Rui YJ, Mi JY. Outcomes of modified trapeziectomy with ligament reconstruction tendon interposition for the treatment of advanced thumb carpometacarpal arthritis: Two-year follow-up. Medicine (Baltimore). 2018 Mar;97(13):e0235. doi: 10.1097/MD.0000000000010235. PMID 29595674
- [Background] Robles-Molina MJ, Lopez-Caba F, Gomez-Sanchez RC, Cardenas-Grande E, Pajares-Lopez M, Hernandez-Cortes P. Trapeziectomy With Ligament Reconstruction and Tendon Interposition Versus a Trapeziometacarpal Prosthesis for the Treatment of Thumb Basal Joint Osteoarthritis. Orthopedics. 2017 Jul 1;40(4):e681-e686. doi: 10.3928/01477447-20170503-03. Epub 2017 May 8. PMID 28481387
- [Background] Degeorge B, Dagneaux L, Andrin J, Lazerges C, Coulet B, Chammas M. Do trapeziometacarpal prosthesis provide better metacarpophalangeal stability than trapeziectomy and ligamentoplasty? Orthop Traumatol Surg Res. 2018 Nov;104(7):1095-1100. doi: 10.1016/j.otsr.2018.07.008. Epub 2018 Aug 11. PMID 30107277
- [Background] Lane JCE, Rodrigues JN, Furniss D, Burn E, Poulter R, Gardiner MD. Basal thumb osteoarthritis surgery improves health state utility irrespective of technique: a study of UK Hand Registry data. J Hand Surg Eur Vol. 2020 Jun;45(5):436-442. doi: 10.1177/1753193420909753. Epub 2020 Mar 12. PMID 32162998
- [Background] Parker S, Riley N, Dean B; Oxford Upper Limb Collaborative. Management of osteoarthritis at the base of the thumb. Bone Joint J. 2020 May;102-B(5):600-605. doi: 10.1302/0301-620X.102B5.BJJ-2019-1464.R2. PMID 32349588
- [Background] Al-Qattan MM, Al Mohrij SA. Mid-Term Results of Partial Trapeziectomy and Simple FCR Tendon Graft Interposition in a Selected Group of Patients with Thumb Carpometacarpal Joint Arthritis. J Hand Microsurg. 2020 Apr;12(1):43-46. doi: 10.1055/s-0039-1698356. Epub 2019 Nov 22. PMID 32280181
- [Background] Shah DS, Middleton C, Gurdezi S, Horwitz MD, Kedgley AE. The Effect of Surgical Treatments for Trapeziometacarpal Osteoarthritis on Wrist Biomechanics: A Cadaver Study. J Hand Surg Am. 2020 May;45(5):389-398. doi: 10.1016/j.jhsa.2019.10.003. Epub 2019 Nov 14. PMID 31733980
- [Background] Chug M, Williams N, Benn D, Brindley S. Outcome of uncemented trapeziometacarpal prosthesis for treatment of thumb carpometacarpal joint arthritis. Indian J Orthop. 2014 Jul;48(4):394-8. doi: 10.4103/0019-5413.136270. PMID 25143644
- [Background] Wajngarten D, Campos JADB, Garcia PPNS. The Disabilities of the Arm, Shoulder and Hand scale in the evaluation of disability - A literature review. Med Lav. 2017 Aug 28;108(4):314-323. doi: 10.23749/mdl.v108i4.6336. PMID 28853432
- [Background] Kroon FPB, Boersma A, Boonen A, van Beest S, Damman W, van der Heijde D, Rosendaal FR, Kloppenburg M. Performance of the Michigan Hand Outcomes Questionnaire in hand osteoarthritis. Osteoarthritis Cartilage. 2018 Dec;26(12):1627-1635. doi: 10.1016/j.joca.2018.07.018. Epub 2018 Aug 9. PMID 30099114
- [Background] Rosales RS, Garcia-Gutierrez R, Reboso-Morales L, Atroshi I. The Spanish version of the Patient-Rated Wrist Evaluation outcome measure: cross-cultural adaptation process, reliability, measurement error and construct validity. Health Qual Life Outcomes. 2017 Aug 24;15(1):169. doi: 10.1186/s12955-017-0745-2. PMID 28836994
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230